CLINICAL TRIAL: NCT05215197
Title: Intracochlear Platelet-rich Fibrin Application in Cochlear Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Head of Department of Otolaryngology, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hearing Loss, Sensorineural
Keywords: cochlear implant; platelet rich fibrin
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: open uncontrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intracochlear prf administration group (Experimental): intracochlear prf administration group
  Interventions: Drug: intracochlear platelet rich fibrin administration

INTERVENTIONS:
Drug: intracochlear platelet rich fibrin administration — intracochlear platelet rich fibrin administration during routine cochlear implantation surgery

SUMMARY:
Fibrosis due to surgical trauma is a common problem with cochlear implants. Fibrosis limits the effectiveness of implant and increases the power consumption. Our aim in this study is to benefit from the anti-inflammatory effects of autologous platelet-rich fibrin to reducing the fibrotic cascade.

DETAILED DESCRIPTION:
The most common problem with cochlear implants is that their effectiveness decreases over time and they are not functional enough mainly due to fibrosis.

Our aim in this study is to benefit from the anti-inflammatory effects of autologous platelet-rich fibrin to reducing the fibrotic cascade.

Cochlear implant application will be performed under general anesthesia. After the postauricular incision and mastoidectomy, posterior tympanotomy will find the middle ear and from there the round window, and platelet fibrin prepared with the i-prf technique will be locally applied to the round window during the operation, and then implantation will be performed.

The points where the electrode enters the cochlea will be covered with fascia.

Intraoperative NRT and impedances will be measured on all electrodes in all patients, and NRT and impedance measurements will be repeated in the 1st week, 1st month, 3rd and 6th months postoperatively.

Custom Sound EP 5.0 (5.0.4.136) program provided by Cochlear company will be used for these measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sensorineural hearing loss
* Patients who will have cochlear implant surgery with CI422 electrode

Exclusion Criteria:

* Patients with cochlear abnormality
* Patients with auditory neuropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Electrode Impedance(Ohm) | 1-6 months
  All intra-operative impedance values will be acquired after surgery. They will be repeated in first week, 1, 3 and 6th months

SECONDARY OUTCOMES:
Electrode thresholds(CL) | 1-6 months
  All intra-operative threshold values will be acquired after surgery. They will be repeated in first week, 1, 3 and 6th months

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The metadata will be shared by a public depository.